CLINICAL TRIAL: NCT01092468
Title: Prospective, Randomised, Single-blinded Study : Comparison of Harmonic Scalpel to Conventional Diathermy in Perforator Flap
Brief Title: Comparison of Harmonic Scalpel to Conventional Diathermy in Perforator Flap Elevation for Head and Neck Reconstruction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Man Ki Chung, Assistant professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009-08-063
Record Dates: First submitted 2010-03-08; First posted 2010-03-25 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Cancer
Keywords: cancer; reconstruction; free flap; surgery
MeSH Terms: conditions — Neoplasms | interventions — Diathermy

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Diathermy (Placebo Comparator): Perforator flap elevation using conventional diathermy technique
  Interventions: Procedure: Diathermy
- Harmonic Scalpel (Active Comparator): Perforator flap elevation using Harmonic Scalpel
  Interventions: Procedure: Harmonic Scalpel

INTERVENTIONS:
Procedure: Diathermy — flap dissection with conventional diathermy
  Arms: Diathermy
Procedure: Harmonic Scalpel — flap dissection using harmonic scalpel (FOCUS)
  Arms: Harmonic Scalpel

SUMMARY:
This study is to compare the efficacy of Harmonic Scalpel with conventional diathermy technique in terms of reducing elevation time and perioperative complications of perforator flaps for head and neck reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* head and neck reconstruction with perforator flap
* informed consent from the patient

Exclusion Criteria:

* coagulation problem
* refused to participate

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
flap elevation time: from identification of skin perforator to completion of dissection to main pedicle | 1 hour after completion of flap elevation

SECONDARY OUTCOMES:
intraoperative complications: bleeding, perforator injury (thermal, mechanical) | 1 hour after completion of flap elevation
postoperative drainage amount | 1 week after flap inset
postoperative pain measured by visual analogue scale (VAS) | 1 week after completion of flap elevation

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical center, Seoul, South Korea